CLINICAL TRIAL: NCT05941286
Title: Effect of Continuous Glucose Monitoring System Alerts on Diabetes Management in the Hospital: a Randomised Controlled Trial
Brief Title: Effect of Continuous Glucose Monitoring System Alerts on Diabetes Management in the Hospital
Acronym: SIGNAL
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Shanghai 6th People's Hospital (Other)
Responsible Party: Principal Investigator, Jian Zhou, Principal Investigator, Professor, Chief Physician, Deputy Director, Shanghai 6th People's Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2023061201
Record Dates: First submitted 2023-07-03; First posted 2023-07-12 (Actual); Last update posted 2025-12-23 (Actual); Status verified 2025-09

CONDITIONS: Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (3):
- CGM system with both glucose predictive alerts and threshold alerts on (Experimental): Patients will wear a real-time CGM (The Guardian Connect CGM System with Guardian sensor 3, Medtronic), which provide glucose readings every 5 minutes for up to 7 days. High/low predictive/threshold alerts will be enabled in this group, with low glucose alert set at 3.9 mmol/L and high glucose alert set at 16.7 mmol/L. Notably, predictive threshold alerts are triggered when a high/low glucose value is predicted within the next 15 min. In addition, patients will undergo POC testing at least 4 times per day (usually before meals and bedtime).
  Interventions: Device: CGM system with both glucose predictive alerts and threshold alerts on
- CGM system with only glucose threshold alerts on (Experimental): Patients will wear a real-time CGM (The Guardian Connect CGM System with Guardian sensor 3, Medtronic), which provide glucose readings every 5 minutes for up to 7 days. Only high/low threshold alerts will be enabled in this group, with the same high/low glucose alert set, which is 3.9 mmol/L and 16.7 mmol/L respectively. In addition, patients will undergo POC testing at least 4 times per day (usually before meals and bedtime).
  Interventions: Device: CGM system with only glucose threshold alerts on
- CGM system with glucose alerts off (Active Comparator): Patients will wear a real-time CGM (The Guardian Connect CGM System with Guardian sensor 3, Medtronic), which provide glucose readings every 5 minutes for up to 7 days. High/low predictive/threshold alerts will be off in this group. In addition, patients will undergo POC testing at least 4 times per day (usually before meals and bedtime).
  Interventions: Device: CGM system with glucose alerts off

INTERVENTIONS:
Device: CGM system with both glucose predictive alerts and threshold alerts on — the cloud-based real-time continuous glucose monitoring and management system with both glucose predictive alerts and threshold alerts on
  Arms: CGM system with both glucose predictive alerts and threshold alerts on
Device: CGM system with only glucose threshold alerts on — the cloud-based real-time continuous glucose monitoring and management system with only glucose threshold alerts on
  Arms: CGM system with only glucose threshold alerts on
Device: CGM system with glucose alerts off — the cloud-based real-time continuous glucose monitoring and management system with glucose predictive/threshold alerts off
  Arms: CGM system with glucose alerts off

SUMMARY:
Current continuous glucose monitoring (CGM) devices provide features that alert for current and impending adverse glycemic events.This trial aims to examine whether these glucose alerts provided added benefit on glycemic outcomes in patients with type 1 or 2 diabetes who required intensive insulin therapy during hospitalization.

DETAILED DESCRIPTION:
Glycemic management for patients with diabetes during hospitalization is highly challenging, especially for those requiring intensive insulin therapy. For those patients, hypoglycemia is a common adverse event, which is associated with adverse clinical outcomes. Bedside capillary point-of-care (POC) glucose monitoring is the standard of care to assess glycemic control in the hospital. However, POC glucose testing only provides glucose measurements at specific time points, leading to missed information important for glycemic control. Continuous glucose monitoring (CGM) measures interstitial glucose every 5 min, thus providing a more complete glycemic profile during a 24 h period compared with standard POC glucose testing.

The cloud-based real-time continuous glucose monitoring (RT-CGM) and management system was previously observed to be safe and effective in guiding intensive insulin therapy. Therefore, this CGM intergraded system holds promise for improving glucose control in patients with diabetes during hospitalization. However, it is currently unclear if alerts are the main reason for the better outcome in the RT-CGM groups, or rather the fact that sensor values are available in real-time. Moreover, the current system provided the feature of predictive threshold alerts that could alert before the onset of clinical hypoglycemia or hyperglycemia. Thus, this trial aims to examine whether these glucose alerts provided added benefit on glycemic outcomes in patients with type 1 or 2 diabetes who required intensive insulin therapy during hospitalization.

ELIGIBILITY:
Inclusion Criteria:

1. Males and females ≥ 18 years.
2. Type 1 or type 2 diabetes with suboptimal glucose control requiring hospitalization, as determined by endocrinologists following clinical guidelines.
3. Willingness and ability to comply with the clinical investigation plan.

Exclusion Criteria:

1. significant hyperglycemia or diabetic ketoacidosis requiring continuous intravenous insulin infusion.
2. Female subjects who are pregnant or have a plan of pregnancy at time of enrollment into the study.
3. Current users of real-time glucose monitoring sensors or flash-glucose monitoring.
4. Participants were unable to tolerate tape adhesive around sensor placement area, or with medically documented allergy towards the adhesive (glue) of plasters, or with serious skin diseases (e.g. psoriasis vulgaris, bacterial skin diseases) around sensor placement area.
5. Patients expected to require operation, admission to the ICU and MRI procedures during hospitalization.
6. Mental condition rendering the subject unable to understand the nature, scope, and possible consequences of the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 533 (Actual)
Dates: Start 2024-04-18 (Actual); Primary Completion 2024-12-16 (Actual); Study Completion 2024-12-16 (Actual)

PRIMARY OUTCOMES:
Time in range (3.9~10.0mmol/L, %) | Through study completion (during hospitalization, 5-7 days)
  Percentage of time within glucose level of 3.9-10.0 mmol/L (70-180 mg/dL) measured by CGM.

SECONDARY OUTCOMES:
Time above range (>10.0mmol/L, %) | Through study completion (during hospitalization, 5-7 days)
  Percentage of time above glucose level of 10.0 mmol/L (180 mg/dL) measured by CGM.
Time above range (>13.9mmol/L, %) | Through study completion (during hospitalization, 5-7 days)
  Percentage of time above glucose level of 13.9 mmol/L (250 mg/dL) measured by CGM.
Time below range (<3.9mmol/L, %) | Through study completion (during hospitalization, 5-7 days)
  Percentage of time below glucose level of 3.9 mmol/L (70 mg/dL) measured by CGM.
Time below range (<3.0mmol/L, %) | Through study completion (during hospitalization, 5-7 days)
  Percentage of time below glucose level of 3.0 mmol/L (54 mg/dL) measured by CGM.
Time in range (3.9~7.8mmol/L, %) | Through study completion (during hospitalization, 5-7 days)
  Percentage of time within glucose level of 3.9-7.8 mmol/L (70-140 mg/dL) measured by CGM.
Glycemia risk index (GRI) | Through study completion (during hospitalization, 5-7 days)
  Glycemia risk index (GRI) was calculated according to the following equation: GRI = (3.0×VLow) + (2.4×Low) + (1.6×VHigh) + (0.8×High).
Mean sensor glucose (MSG) | Through study completion (during hospitalization, 5-7 days)
  Mean of daily continuous 24-h blood glucose.
Coefficient of variation (CV) | Through study completion (during hospitalization, 5-7 days)
  Standard deviation divided by mean glucose level measured by CGM.
Standard deviation (SD) | Through study completion (during hospitalization, 5-7 days)
  Standard deviation of blood glucose measurements during CGM.

OTHER OUTCOMES:
Time taken to achieve target glucose (days) | Through study completion (during hospitalization, 5-7 days)
  Target glucose was defined as CGM-recorded TIR 3.9-10.0 mmol/L (70-180 mg/dL) more than 70%, with a maximum allowed time of 7 days.
Length of hospital stay (days) | Through study completion (during hospitalization, 5-7 days)
  The total length of hospital stay.
Total daily insulin dose (units/kg/day) | Through study completion (during hospitalization, 5-7 days)
  Total daily insulin dose per kilogram of body weight per day.
Total daily basal insulin dose (units/kg/day) | Through study completion (during hospitalization, 5-7 days)
  Total daily basal insulin dose per kilogram of body weight per day.
Total prandial insulin dose (units/kg/day) | Through study completion (during hospitalization, 5-7 days)
  Total prandial basal insulin dose per kilogram of body weight per day.

CONTACTS AND LOCATIONS:
Overall Officials: Jian Zhou, Principal Investigator — Shanghai 6th People's Hospital
Locations (1):
- Shanghai Sixth People's Hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No